CLINICAL TRIAL: NCT03257254
Title: Observational Study of the Effect of VarIthena® on Wound Healing in the Treatment of Venous Leg Ulcers Resulting From Chronic Venous Insufficiency
Brief Title: Effect of VarIthena on Wound Healing in Venous Leg Ulcers (VLU)
Acronym: VIEW-VLU
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: BTG-001652-01
Record Dates: First submitted 2017-08-16; First posted 2017-08-22 (Actual); Results first posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Venous Leg Ulcer
Keywords: GSV; AASV; Vein; Venous; Ulcer; Varicose Vein; VLU; venous insufficiency; venous disease; chronic VLU
MeSH Terms: conditions — Varicose Ulcer; Ulcer; Varicose Veins; Venous Insufficiency | interventions — Polidocanol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Varithena — Administration procedures and volume are per standard of care, full prescribing information, and instructions for use.

SUMMARY:
A 12 month, multicenter, open-label registry to observe chronic venous insufficiency resulting in VLU treated with Varithena.

DETAILED DESCRIPTION:
This 12 month, multicenter, open-label registry is designed to collect treatment and outcome data related to participants treated with Varithena for great saphenous vein (GSV) system and/or anterior accessory saphenous vein (AASV) incompetence resulting in VLU. Participant are treated per Investigator's Standard of Care (SoC) and in accordance with the Full Prescribing Information (FPI) and Instructions for Use (IFU). For participants with healed ulcers during the 12 month follow-up period, VLU recurrence information is collected.

ELIGIBILITY:
Inclusion Criteria:

* Men and women; age ≥18
* Investigator has selected Varithena® to treat participants classified C6 with chronic (≥3 months) VLU resulting from GSV and/or AASV incompetence
* Wound can be visualized in one plane to allow for image collection of the entire wound in one photograph, or if wound is circumferential, participant must be able to capture the entire wound using multiple photographs taken from directly above the wound (straight on)
* Reflux >500 milliseconds (ms) on duplex ultrasound
* Willing and able to collect wound photographs and data using an application installed on a tablet
* Willing and able to return for scheduled follow-up and wound care visits
* Ability to comprehend and sign informed consent form (ICF) and complete questionnaires

Exclusion Criteria:

* Contraindications to Varithena® 1% in accordance with the FPI
* Any serious concomitant disease, per physician's discretion, that confounds wound healing, including malignant changes of wound
* Concomitant heat ablation, or heat ablation of index leg within 6 weeks prior to treatment with Varithena®
* Significant arterial disease or ankle-brachial pressure index (ABPI) ≤0.8
* In the opinion of Investigator, wound would close within 12 weeks without additional treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants classified C6 on Clinical-Etiology-Anatomy-Pathophysiology (CEAP) classification with active VLU resulting from venous insufficiency of the GSV system and/or AASV
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shao, MD, Principal Investigator — Swedish Covenant Hospital
Locations (14):
- United States (13):
  - Stanford University, Palo Alto, California
  - University of California Davis Health, Sacramento, California
  - The Vascular Experts, Darien, Connecticut
  - Pines Clinical Research, Aventura, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Swedish Covenant Hospital, Chicago, Illinois
  - Mass General, Boston, Boston, Massachusetts
  - The Venous Institute of Buffalo, Buffalo, New York
  - Mercy Health Cincinnati -West Hospital, Cincinnati, Ohio
  - OhioHealth Research, Columbus, Ohio
  - Totality, Oklahoma City, Oklahoma
  - University of Texas Health Sciences Center at Houston, Houston, Texas
  - Lake Washington Vascular, PLLC, Bellevue, Washington
- Oakville Vascular, Oakville, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Prospective Registry Cohort: Participants classified C6 on Clinical-Etiology-Anatomy-Pathophysiology (CEAP) classification with active VLU resulting from venous insufficiency of the GSV system and/or AASV treated with Varithena.
Period: Overall Study
Arm/Group | Prospective Registry Cohort
Started | 76
Completed | 55
Not Completed | 21
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 9
Not completed — Study discontinued by sponsor | 5

BASELINE CHARACTERISTICS:
Arm/Group | Prospective Registry Cohort
Number analyzed (Participants) | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 9
  United States | 67

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Wound Perimeter
Description: Mean change in wound perimeter as measured by photograph inputted into wound measuring technology platform. Larger number indicates a lower wound perimeter compared to baseline. Epithelial migration measured by change in perimeter of wound.
Time Frame: Baseline to 12 weeks and to 12 months
Population: Based on number of wounds continuing to heal at the timepoint.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: wounds
Arm/Group | Prospective Registry Cohort
Number analyzed (Participants) | 76
Number analyzed (wounds) | 80
mm
  at 12 weeks | 29.36 (146.13)
  at 12 months | 43.64 (2.6)

2. Primary Outcome: Number of Wound Closure at 12 Weeks
Description: Total number of healed wounds at 12 weeks post treatment. Wound healing is measured measured by photograph inputted into wound measuring technology platform.
Time Frame: Baseline to 12 weeks
Measure: Number; unit: wounds
Units Other Than Participants: wounds
Arm/Group | Prospective Registry Cohort
Number analyzed (Participants) | 76
Number analyzed (wounds) | 80
wounds | 43

3. Primary Outcome: Time to Wound Closure
Description: Median number of days to wound closure measured weekly. Wound closure as measured by photograph inputted into wound measuring technology platform.
Time Frame: Baseline to wound closure or to 12 months, whichever occurs first
Measure: Median (95% Confidence Interval); unit: days
Units Other Than Participants: wounds
Arm/Group | Prospective Registry Cohort
Number analyzed (Participants) | 76
Number analyzed (wounds) | 80
days | 89 [62 to 117]

4. Secondary Outcome: Change in Pain
Description: Mean change in pain on numeric pain rating scale (NPRS) compared to baseline at 12 months post-treatment. Minimum value is "0" and maximum value is "10". Higher scores mean a worse outcome.
Time Frame: Baseline to 12 weeks and to 12 months
Population: Analysis is based on the number of wounds and not number of patients. If a patient had more than one reported pain score during a timepoint, the worst (highest) NPRS score was used for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: wounds
Arm/Group | Prospective Registry Cohort
Number analyzed (Participants) | 76
Number analyzed (wounds) | 80
score on a scale
  at 12 weeks | -1.4 (3.1)
  at 12 months | -2.5 (3.1)

5. Secondary Outcome: Change on EQ-5D-5L Quality of Life Assessment
Description: Mean change on 5-level EQ-5D (EQ-5D-5L) quality of life assessment compared to baseline at 12 months post-treatment. Minimum value is "0" and maximum value is "1". Higher score mean better outcome.
Time Frame: Baseline to 12 weeks and to 12 months
Population: Statistics are based on the number of wounds and not number of patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: wounds
Arm/Group | Prospective Registry Cohort
Number analyzed (Participants) | 76
Number analyzed (wounds) | 80
score on a scale
  at 12 weeks | 0.066 (0.233)
  at 12 months | 0.072 (0.223)

6. Secondary Outcome: Change in VCSS
Description: Mean change in Venous Clinical Severity Score (VCSS) from baseline to 12 month follow up. VCSS assesses nine common signs/symptoms of venous disease and each item is scored individually with a minimum score of "0" and maximum score of "3". The individual items are added together to assess change from baseline. Higher scores mean worst outcome.
Time Frame: Baseline to 12 weeks and to 12 months
Population: Analysis is based on number of wounds and not number of patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: wounds
Arm/Group | Prospective Registry Cohort
Number analyzed (Participants) | 76
Number analyzed (wounds) | 80
score on a scale
  at 12 weeks | -5.8 (5.6)
  at 12 months | -10.0 (7.1)

7. Secondary Outcome: Number of Wounds Remaining Closed at 3 Months Post-wound Closure Date
Description: Count of wounds remaining closed at 3 months post-wound closure determined via photograph and assessed by wound measurement technology platform.
Time Frame: Baseline to 12 months
Population: 54 wounds were closed prior to the 12-month follow up visit.
Measure: Count of Units; unit: wounds
Units Other Than Participants: wounds
Arm/Group | Prospective Registry Cohort
Number analyzed (Participants) | 76
Number analyzed (wounds) | 54
wounds | 47

8. Secondary Outcome: Number of Wound Recurrences
Description: Count of wound recurrences of healed wounds. For healed wounds, VLU recurrence was collected via phone calls and subjects at follow up timelines.
Time Frame: Baseline to 12 months
Population: 54 wounds were closed prior to the 12 month follow up.
Measure: Number (95% Confidence Interval); unit: wounds
Units Other Than Participants: wounds
Arm/Group | Prospective Registry Cohort
Number analyzed (Participants) | 76
Number analyzed (wounds) | 54
wounds | 7 [5.4 to 24.9]

9. Secondary Outcome: Number of Ulcer Free Days
Description: Mean number of ulcer free days defined as days from baseline to date of recurrence
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Prospective Registry Cohort
Number analyzed (Participants) | 76
days | 240.5 (118.9)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during a 1 year period starting from the initiation of treatment until the subject completes the registry follow up period or withdraws.
Arm/Group | Prospective Registry Cohort
All-Cause Mortality (participants affected / at risk) | 0/76
Serious Adverse Events (participants affected / at risk) | 6/76
Other Adverse Events (participants affected / at risk) | 1/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prospective Registry Cohort (N=76)
Peripheral arterial occlusive disease (Vascular disorders) | 1
Asthenia (General disorders) | 1
Staphylococcal infection (Infections and infestations) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Sepsis (Infections and infestations) | 2
Polyarteritis nodosa (Vascular disorders) | 1
Gangrene (Vascular disorders) | 1
Cellulitis (Infections and infestations) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Toe amputation (Surgical and medical procedures) | 1
Condition aggravated (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prospective Registry Cohort (N=76)
Blister (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/54/NCT03257254/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT03257254/SAP_001.pdf